CLINICAL TRIAL: NCT04618068
Title: Prevalence of Different Stages of Periodontal Diseases Among a Sample of Young Adult Obese Egyptian Patients: A Hospital Based Cross-Sectional Study
Brief Title: Prevalence of Periodontal Diseases Among Obese Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yasmine Abbas Elsayed (Other)
Responsible Party: Sponsor-Investigator, Yasmine Abbas Elsayed, master postgraduate student, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 21252462
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is a cross-sectional survey investigating the Prevalence of Different Stages of Periodontal Diseases among a sample of Young Adult Obese Egyptian patients attending the oral diagnosis clinic at faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
In recent years, research has focused on the relationship between periodontitis and systemic disorders such as diabetes mellitus, rheumatoid arthritis, cardiovascular diseases and obesity. Obesity is the result of many disorders arising from several different causes, including complex interactions among genetic, biochemical, neural and psychological factors as well as environmental, social and economic factors. Moreover, obesity is considered itself a risk factor for several diseases, such as type 2 diabetes mellitus, cardiovascular disease, tumors and potentially for periodontal disease.

Obesity has a significant association with periodontitis in terms of body mass index (BMI), waist-to-hip circumference ratio, body fat, and maximum oxygen consumption. The BMI has always been considered a simple method for analysis of the nutritional status by world health organization. In 2014, the world health organization (WHO) estimated that around 600 million obese adults worldwide were obese and a further increase is expected in the future due to increased consumption of high-calorie diets and a sedentary lifestyle.

A bidirectional relationship links metabolic disorders like type 2 diabetes or obesity and periodontitis The common soil between these chronic conditions is likely to be systemic, low-grade inflammation: dental plaque releases bioactive products, which in turn stimulate host responses at the gingival and systemic level, promoting the release of inflammatory cytokines. These mediators are implicated in insulin resistance, impaired β-cell function, endothelial dysfunction, driving diabetes onset and the accelerating atherosclerosis marking it.

The association between obesity and periodontitis is one of the most recent fields of research in periodontal medicine and the possible underlying biological mechanisms remain unclear. Since then, the hypothesis that obesity is a risk factor for periodontitis has been evidenced by several epidemiological studies. The visceral adipose tissue has been shown to act as an organ that secretes important bioactive substances termed adipocytokines, including tumor necrosis factor alpha, which may affect periodontal disease pathogenesis

A recent study has shown that in a population young adults, tumor necrosis factor levels in gingival crevicular fluid correlate with individuals with BMI greater than forty. The authors suggested that obesity is type of low grade systemic inflammatory disease affecting periodontal disease progression. The systemic inflammation associated with obesity may increase susceptibility to chronic infectious diseases, which may explain how obesity would affect the development of periodontal diseases. However, whether obesity and overweight are associated with periodontitis is still under debate.

Many clinical studies have shown that overweight status, obesity, weight gain, and increased waist circumference are risk factors for the development of periodontitis or the worsening of periodontal status. Patients presenting moderate and severe periodontal disease have been found to produce higher systemic levels of inflammatory and immune markers. Treatment of periodontal disease can reduce these markers. Since the first report suggesting in a rat models existence of a possible relation between obesity and periodontal disease in 1977, only 21 years later, the first human study on the Japanese population, revealing that obese subjects showed a probability of suffering from periodontitis 8.6 times greater than non-obese ones.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is between 18-39 years old as the strength and physical performance reach their peak from 18-39 years
2. Body mass index more than 30.
3. Patient consulting in the outpatient clinic.
4. Provide informed consent.

Exclusion Criteria:

1. Patients who have a systemic disease or were on medication for any systemic disease/conditions.
2. Patients who received periodontal treatment or antibiotics for at least 3 months.
3. Completely edentulous or having removable prosthetic appliance.
4. Pregnant women or lactating mothers.
5. Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University. Medical history will be taken, thorough oral examination will be done, and a full questionnaire will be filled for each patient.
  The questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions. It will include a section for demographic information of age, sex, social and educational of the patient. It will include questions about medical condition, habits of trauma, smoking and its frequency.
Sampling Method: Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The prevalence of periodontal disease in obese Egyptian patients | after recruitment of required sample size , through study completion an average of one year
  we need to know the prevalence of periodontal disease in obese Egyptian patients

CONTACTS AND LOCATIONS:
Overall Officials: Noha Ayman Ghallab, Professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry , Cairo Univeristy, Cairo, Egypt

REFERENCES:
- [Derived] Abbas Y, Elsaadany B, Ghallab N. Prevalence of different stages of periodontal diseases among a sample of young adult obese Egyptian patients: a hospital based Cross-sectional study over 1 year. BMC Oral Health. 2023 Aug 16;23(1):573. doi: 10.1186/s12903-023-03278-3. PMID 37582775